CLINICAL TRIAL: NCT01615458
Title: Disseminating Evidence-based Mood Disorder Chronic Care Models
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Amy M. Kilbourne, Associate Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: G009567
Record Dates: First submitted 2012-06-06; First posted 2012-06-08 (Estimated); Last update posted 2012-06-11 (Estimated); Status verified 2012-06

CONDITIONS: Bipolar Disorder; Depression
Keywords: Care Management; Implementation; Intervention; Mood Disorders
MeSH Terms: conditions — Bipolar Disorder; Depression; Mood Disorders | interventions — Chronic Care Model

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Usual Care (Active Comparator): Patients will receive their usual care from providers at the clinic.
  Interventions: Behavioral: Chronic Care Model for Mood Disorders

INTERVENTIONS:
Behavioral: Chronic Care Model for Mood Disorders — CCM includes (1) patient self-management enhancement focused on promoting healthy lifestyles as coping strategies to minimize the negative impact of depressive, manic, and other affective symptoms; (2) provider support for evidence-based decision-making; and (3) enhanced access and continuity for anticipatory rather than reactive care.
  Other Names: Life Goals Collaborative Care

SUMMARY:
This study will determine if a version of the chronic care model for individuals with mood disorders can improve patient health.

DETAILED DESCRIPTION:
Chronic mood disorders (notably, bipolar disorder and recurrent unipolar major depressive disorder) are associated with substantial functional impairment, morbidity, economic burden, and mortality. Depression and bipolar disorder are common and are the leading causes of disability worldwide, are associated with substantial costs, and when left untreated, can lead to premature mortality, particularly from suicide. Despite the proliferation of evidence-based guidelines for the treatment of mood disorders, the quality of care and subsequent outcomes remain suboptimal for those suffering from these illnesses.

Collaborative chronic care models (CCMs) have demonstrated efficacy and cost-effectiveness in managing depression and more recently, bipolar disorder. Many of the successful interventions to improve depression treatment and outcomes (e.g., PROSPECT) are based on the Chronic Care Model (CCM). These treatment models combine patient self-management education with ongoing care coordination that is delivered by a care manager, who coordinates care with primary care and mental health providers and facilitates systematic dissemination of guidelines related to mood disorders treatment. In bipolar disorder, CCMs have been found to be cost-neutral, and in depression, cost-effective compared to usual care; hence making business cases for CCMs is promising in both the private and public sectors.

There is mounting demand for CCMs to be implemented for patients across different mental health diagnoses, in order to maximize their reach across diverse clinic populations, and to make them more appealing to healthcare providers, who might be reluctant to hire multiple care managers for different conditions. Unipolar major depressive and bipolar disorders are some of the most common forms of mood disorders treated in specialty mental health as well as in primary care settings. Up to 5.5% and 16.2% of the population have bipolar spectrum disorder and unipolar major depressive disorder, respectively. Based on pilot data from Colorado Access, about a third of patents being treated for depression in routine care settings screened positive for bipolar disorder. Moreover, only a third of patients with unipolar depression remit, which in part might be attributed to under-treatment or inappropriate treatment of bipolar II disorder. However, while CCMs for unipolar depression and bipolar disorder exist, to date they have not been implemented in combination. This project will pilot test a combined CCM that can be applied to patients with unipolar depression or bipolar disorder in specialty mental health or primary care clinics.

This is a one-year pilot randomized controlled trial comparing LGCC to usual care that will involve patients diagnosed with bipolar disorder or unipolar depression who are receiving care in clinics affiliated with NNDC sites or unaffiliated primary care sites. The project will be implemented in three phases: training of existing staff at the local Depression Center clinics, implementation of LGCC, and final outcomes evaluation to inform future studies. Patients from up to four mental health clinics affiliated with NNDC sites (University of Michigan Depression Center, Stanford University Depression Center, University of Colorado-Denver Depression Center, and University of California-San Francisco Depression Center) and 1 primary care setting (Packard Community Health, Ann Arbor, MI) will be randomized to receive LGCC or standard care as usual (32 per site; total 160 patients). Randomization will be stratified by diagnosis (unipolar depression or bipolar disorder). At the end of the pilot study, patients not randomized to receive LGCC will be offered the intervention. An additional 10 providers will be asked to complete surveys from their site (total n=50), for a grand total of n=210 participants (160 patients and 50 providers).

ELIGIBILITY:
Inclusion Criteria:

* Currently being seen as a patient at the participating site
* Active diagnosis or treatment plan for Bipolar Disorder (I, II, NOS) or unipolar depression.

Exclusion Criteria:

* No active substance intoxication
* No acute medical illness or dementia
* No active suicidal ideation at time of participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-07; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Quality of Life | Change in From Baseline in Quality of Life at 6-months.
Decreased Mood Disorder Symptoms | Change from Baseline in Mood Disorder Symptoms at 6-months

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Stanford University, Palo Alto, California
  - University of California- San Francisco, San Francisco, California
  - University of Colorado- Denver, Denver, Colorado
  - University of Michigan, Ann Arbor, Michigan